CLINICAL TRIAL: NCT01714427
Title: Validation of a Lung Inflammation Model in Healthy Volunteers by Radiological Tools and Glucocorticoid Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernd Jilma, Associate Professor of Clinical Pharmacology & Internal Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DEXA - LIM
Record Dates: First submitted 2011-09-06; First posted 2012-10-26 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Experimental Lung Inflammation
MeSH Terms: conditions — Pneumonia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Sterile isotonic saline (Placebo Comparator)
  Interventions: Drug: Sterile isotonic saline

INTERVENTIONS:
Drug: Dexamethasone — Two doses of 40mg dexamethasone (in 100 ml physiologic saline solution, respectively) will be administered intravenously prior to LPS instillation.
  Arms: Dexamethasone
Drug: Sterile isotonic saline — two doses of 100 ml physiologic saline solution will be administered intravenously prior to LPS instillation.
  Arms: Sterile isotonic saline

SUMMARY:
The purpose of this study is to investigate the local and systemic inflammatory response and haemostatic alterations in the lungs after lipopolysaccharide (LPS) instillation and to determine the feasibility of imaging techniques to quantify lung inflammation in an adapted human endotoxin instillation model.

The investigators will also explore whether glucocorticoid treatment can blunt LPS effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities. (Trial activities are any procedure that would not have been performed during normal management of the subject).
* Nonsmoker
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* If female and of childbearing potential and subjects agrees to employ adequate birth control measures (e. g. oral contraceptives, barrier method)
* Negative urine pregnancy test

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Pregnancy or Lactation
* Treatment with an investigational drug within three weeks prior to this trial
* Participation in an LPS trial within the last 6 weeks
* Smoking
* History of relevant cardiac arrhythmia
* Preexisting open or closed angle glaucoma
* History of Osteoporosis, Cushing´s syndrome, gastro-duodenal ulcera, cardiovascular disease, vasculitis, diabetes mellitus, hypertension, brain tumor or history of neurosurgery
* Systemic tuberculosis
* Hemorrhagic diathesis
* Relevant liver or kidney dysfunction
* Regular use of medication or abuse of alcohol unless considered clinically relevant
* Use of any medication within one week prior to the first trial day
* Symptoms of a clinically relevant illness in the 3 weeks before the first trial day
* Excessive sporting activities
* Rosacea
* Subjects on Monoamine oxidase inhibitors (should be stopped for at least two to three weeks before dihydrocodeine treatment is initiate)
* Known acute or active hepatic disease within the past 3 months
* A platelet count < 100,000 x 106/L, prothrombin time > 1.5, liver enzymes> 3 times the upper normal limit
* Having received a vaccination up to 8 weeks before the trial

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The effects of LPS instillation on a putative microvascular leak formation in a lung subsegment by radiologic imaging (magnetic resonance imaging, computed tomography) will be quantified. | 6/24 hours after LPS Instillation

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna, Waehringerguertel 18-20, A-1090 Vienna, Austria
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria